CLINICAL TRIAL: NCT03442699
Title: An Initial Feasibility Study of Brief Cognitive Behavioral Therapy for Suicidal Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, David Tolin, Director, Anxiety Disorders Center, Hartford Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHC-2017-0218
Record Dates: First submitted 2018-01-30; First posted 2018-02-22 (Actual); Results first posted 2019-12-30 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Suicide, Attempted
Keywords: cognitive behavioral therapy; suicidal ideology; suicidal behavior
MeSH Terms: conditions — Suicide, Attempted | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will receive up to 10 daily sessions of CBT (depending on length of stay), for about an hour each day. During this time the therapist will work with participants to develop a crisis response plan and build coping skills to prevent future suicidal thoughts and behaviors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy (Experimental): Participants will receive up to 10 daily sessions of cognitive behavioral therapy (depending on length of stay), for about an hour each day. During this time the therapist will work to develop a crisis response plan and build coping skills to prevent future suicidal thoughts and behaviors.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Up to 10 daily sessions of brief cognitive behavioral therapy for suicidal inpatients for about an hour each day.

SUMMARY:
Suicide is a major public health problem. Although inpatient treatment provides immediate stabilization and crisis management, the risk of suicide post-discharge is substantial. Approximately one third of all suicides by individuals with mental disorders occur in the 90 days following hospitalization. Cognitive behavioral therapy (CBT) has been shown to reduce both suicidal ideation and behavior in outpatients. However, to date, the efficacy of inpatient CBT for suicide prevention is not clear. This study aims to 1) develop and implement a brief CBT treatment for suicide prevention for inpatients, 2) conduct a brief feasibility test and collect initial pilot data on efficacy, and 3) collect preliminary data on the effects of CBT on implicit cognitive suicide associations. In Phase 1, the investigators will work with an expert in CBT for suicide prevention to modify his treatment protocol for use with inpatients, and meet with this expert for a 2-day protocol training. In Phase 2, the investigators will conduct an initial feasibility trial with 5-10 inpatients recruited from the Institute of Living inpatient units. Participants will be recruited within 24 hrs of admission or later and will provide written informed consent prior to any study procedures. Enrolled participants will undergo a clinical assessment by an independent evaluator (IE) that will include diagnostic/symptom assessments, assessment of suicide risk using the Columbia-Suicide Rating Scale, and an implicit association test (IAT). Participants will receive up to 10 daily sessions of CBT (depending on length of stay), lasting 1 hour, following the manualized protocol developed in Phase 1. Participants will then meet with the IE again for reassessment after the 10th session or within 24 hr prior to discharge, whichever comes first. After discharge, participants will have a telephone interview at 1 month, 2 month, and 3 month follow-up. The IE will administer the C-SSRS during these calls. The proposed study will yield feasibility and initial efficacy data that will be used to inform a grant proposal to the American Foundation for Suicide Prevention. That proposal will fund a randomized controlled trial of CBT vs. treatment as usual. Concurrently, the investigators will develop an in-house program to train other staff in the protocol, and will submit a second grant to investigate the efficacy of the training program as well as the efficacy of CBT by those clinicians.

DETAILED DESCRIPTION:
Rationale. Suicide is a major public health problem: suicidal ideation affects 14% of the adult U.S. population, and as many as 5% have a lifetime history of suicide attempts.1 Among individuals with depressive disorders, there is an 11% mortality rate from suicide.2 Although inpatient treatment provides immediate stabilization and crisis management, the risk of suicide post-discharge is substantial. Approximately one third of all suicides by individuals with mental disorders occur in the 90 days following hospitalization.3 A review of nearly 2 million adult psychiatric inpatients found that the suicide rate in the 90 days after discharge for patients diagnosed with depressive disorders was 235.1 per 100,000 person-years, markedly higher than that in the US general population (14.2 per 100,000 person-years).4

Cognitive behavioral therapy (CBT) has been shown to reduce both suicidal ideation and behavior.5-8 Though specific protocols vary, typical interventions include problem-solving training,9 cognitive restructuring,10 and training in emotion regulation skills.11 To date, most of the existing research on CBT has been in outpatient samples, and the efficacy of inpatient CBT for suicide prevention is not clear.

Project Aims. The aims of the proposed project are to:

1. develop and implement a brief CBT for suicide prevention on the adult inpatient units;
2. conduct a brief feasibility test and collect initial pilot data on efficacy; and
3. collect preliminary data on the effects of CBT on implicit cognitive suicide associations.

Method. The investigators selected Rudd et al.'s12 CBT protocol for the proposed project. This protocol was tested in a randomized controlled trial (RCT) of outpatients and resulted in a significant reduction in suicide attempts over a 24-month follow-up assessment (hazard ratio = 0.38); those receiving CBT were 60% less likely to make a suicide attempt than were those receiving treatment as usual.13 Of the 6 RCTs that measured suicidal behavior, this was the strongest behavioral effect documented.7

There will be two phases involved in this project, which are described below:

In Phase 1 of the project, the investigators will work with Dr. Rudd to modify his treatment protocol for use in an inpatient setting, and attend a two-day training in the protocol from Dr. Rudd.

In Phase 2 of the project, the investigators will conduct an initial feasibility trial with 5-10 inpatients.

Participants. The investigators will recruit 5-10 consecutive adult inpatients (dependent on flow within the 6-month treatment window) from the Donnelly units.

Procedures. It is anticipated that the treatment component of the study will take place over a period of six months.

Participants will be recruited by a member of the research staff on the day following their inpatient admission or later (for example in the case of a Saturday admission). Patients who meet all of the inclusion criteria and none of the exclusion criteria and agree to participate will provide written informed consent prior to any study procedures. Informed consent will be documented using the Documentation of Informed Consent Form. For patients who are admitted to the hospital involuntarily documentation of competency to provide consent will be completed as well. Only those involuntarily committed patients who have been found competent to provide informed consent for research will be consented. Patients who decline participation will not be approached again. Patients who agree to participation will undergo the informed consent process. This process will involve providing the patient with the informed consent and HIPAA authorization forms to read. The study staff member obtaining consent will highlight the voluntary nature of the research and emphasize that the patient's decision whether or not to participate will not impact his "usual care" treatment plan; however, patients will also be informed that the information discussed with the study clinician is shared with the inpatient treatment team, and thus may be used by them when making decisions about discharge planning. Patients will be informed that they may keep the forms to review with others if they wish to do so before signing. In addition, all questions the patient has about study participation will be answered prior to obtaining written consent.

Enrolled participants will undergo a clinical assessment by an independent evaluator (IE), who will administer the DIAMOND, C-SSRS, SIGH-D, and IAT.

Participants will receive up to 10 daily sessions of CBT (depending on length of stay), lasting 1.5 hours for the first session and 1 hour for the remaining sessions, following the manualized protocol developed in Phase 1. The CBT protocol is designed to be delivered in two phases. In phase I, the therapist conducts a detailed assessment of the patient's most recent suicidal episode or suicide attempt, identifies patient-specific factors that contribute to and maintain suicidal behaviors, provides a cognitive behavioral conceptualization, collaboratively develops a crisis response plan. The crisis response plan is reviewed and updated in each session by adding new skills and/or removing skills determined to be ineffective, impractical, or too challenging. In phase II, the therapist teaches the patient new coping skills inclusion emotion regulation strategies (e.g., relaxation, mindfulness) and cognitive strategies to reduce beliefs and assumptions that serve as vulnerabilities to suicidal behavior (e.g., hopelessness, perceived burdensomeness, guilt and shame). During the first session of CBT, participants are provided with a small pocket-sized notebook (called a "smart book") in which they are directed to record a "lesson learned" at the conclusion of each session. Lessons learned include new skills learned or knowledge gained by participants during each session. Participants are encouraged to use the smart book in the future as a memory aid for managing emotional distress and solving problems.

Participants will then meet with the IE again for the C-SSRS, SIGH-D, IAT, and CSQ after the 10th session or within 24 hrs. prior to discharge, whichever comes first. After discharge, participants will have a telephone interview at 1 month, 2 month, and 3 month follow-up. The IE will administer the C-SSRS during these calls.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* age 18-65 inclusive
* fluent in English (speaking, reading, and writing)
* having made a suicide attempt within one week preceding admission. Admission will be defined as admission to either Hartford Hospital medical floor (in cases where medical stabilization is required prior to transfer to IOL) or to IOL (in cases where medical stabilization is not required). A suicide attempt will be defined as behavior that is self-directed and deliberately results in injury or the potential for injury to oneself for which there is evidence, whether explicit or implicit, of intent to die.

Exclusion Criteria:

* age <18 or ≥66 years old
* history of schizophrenia spectrum disorder
* history of mental retardation or organic brain illness
* current substance use disorder
* active mania or other psychiatric or medical condition that would preclude informed consent or participation in the trial, in the investigator's opinion
* ECT included on patient's inpatient treatment plan. Patients who are referred for ECT after starting the study will be withdrawn from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Tolin, Ph.D., Principal Investigator — Institute of Living/Hartford Hospital
Locations (1):
- Institute of Living, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Borges G, Walters EE. Prevalence of and risk factors for lifetime suicide attempts in the National Comorbidity Survey. Arch Gen Psychiatry. 1999 Jul;56(7):617-26. doi: 10.1001/archpsyc.56.7.617. PMID 10401507
- [Background] Wulsin LR, Vaillant GE, Wells VE. A systematic review of the mortality of depression. Psychosom Med. 1999 Jan-Feb;61(1):6-17. doi: 10.1097/00006842-199901000-00003. PMID 10024062
- [Background] Huisman A, Kerkhof AJ, Robben PB. Suicides in users of mental health care services: treatment characteristics and hindsight reflections. Suicide Life Threat Behav. 2011 Feb;41(1):41-9. doi: 10.1111/j.1943-278X.2010.00015.x. PMID 21309823
- [Background] Olfson M, Wall M, Wang S, Crystal S, Liu SM, Gerhard T, Blanco C. Short-term Suicide Risk After Psychiatric Hospital Discharge. JAMA Psychiatry. 2016 Nov 1;73(11):1119-1126. doi: 10.1001/jamapsychiatry.2016.2035. PMID 27654151
- [Background] Tarrier N, Taylor K, Gooding P. Cognitive-behavioral interventions to reduce suicide behavior: a systematic review and meta-analysis. Behav Modif. 2008 Jan;32(1):77-108. doi: 10.1177/0145445507304728. PMID 18096973
- [Background] Mann JJ, Apter A, Bertolote J, Beautrais A, Currier D, Haas A, Hegerl U, Lonnqvist J, Malone K, Marusic A, Mehlum L, Patton G, Phillips M, Rutz W, Rihmer Z, Schmidtke A, Shaffer D, Silverman M, Takahashi Y, Varnik A, Wasserman D, Yip P, Hendin H. Suicide prevention strategies: a systematic review. JAMA. 2005 Oct 26;294(16):2064-74. doi: 10.1001/jama.294.16.2064. PMID 16249421
- [Background] Mewton L, Andrews G. Cognitive behavioral therapy for suicidal behaviors: improving patient outcomes. Psychol Res Behav Manag. 2016 Mar 3;9:21-9. doi: 10.2147/PRBM.S84589. eCollection 2016. PMID 27042148
- [Background] Hepp U, Wittmann L, Schnyder U, Michel K. Psychological and psychosocial interventions after attempted suicide: an overview of treatment studies. Crisis. 2004;25(3):108-17. doi: 10.1027/0227-5910.25.3.108. PMID 15387237
- [Background] Salkovskis PM, Atha C, Storer D. Cognitive-behavioural problem solving in the treatment of patients who repeatedly attempt suicide. A controlled trial. Br J Psychiatry. 1990 Dec;157:871-6. doi: 10.1192/bjp.157.6.871. PMID 2289097
- [Background] Brown GK, Ten Have T, Henriques GR, Xie SX, Hollander JE, Beck AT. Cognitive therapy for the prevention of suicide attempts: a randomized controlled trial. JAMA. 2005 Aug 3;294(5):563-70. doi: 10.1001/jama.294.5.563. PMID 16077050
- [Background] Linehan MM, Armstrong HE, Suarez A, Allmon D, Heard HL. Cognitive-behavioral treatment of chronically parasuicidal borderline patients. Arch Gen Psychiatry. 1991 Dec;48(12):1060-4. doi: 10.1001/archpsyc.1991.01810360024003. PMID 1845222
- [Background] Rudd MD, Joiner TE, Rajab MH. Treating suicidal behavior: An effective, time-limited approach. New York: Guilford Press; 2001.
- [Background] Rudd MD, Bryan CJ, Wertenberger EG, Peterson AL, Young-McCaughan S, Mintz J, Williams SR, Arne KA, Breitbach J, Delano K, Wilkinson E, Bruce TO. Brief cognitive-behavioral therapy effects on post-treatment suicide attempts in a military sample: results of a randomized clinical trial with 2-year follow-up. Am J Psychiatry. 2015 May;172(5):441-9. doi: 10.1176/appi.ajp.2014.14070843. Epub 2015 Feb 13. PMID 25677353
- [Background] Tolin DF, Gilliam C, Wootton BM, Bowe W, Bragdon LB, Davis E, Hannan SE, Steinman SA, Worden B, Hallion LS. Psychometric Properties of a Structured Diagnostic Interview for DSM-5 Anxiety, Mood, and Obsessive-Compulsive and Related Disorders. Assessment. 2018 Jan;25(1):3-13. doi: 10.1177/1073191116638410. Epub 2016 Mar 17. PMID 26988404
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Williams JB. A structured interview guide for the Hamilton Depression Rating Scale. Arch Gen Psychiatry. 1988 Aug;45(8):742-7. doi: 10.1001/archpsyc.1988.01800320058007. PMID 3395203
- [Background] Borkovec TD, Nau SD. Credibility of analogue therapy rationales. J. Behav. Ther. Exp. Psychiatry. 1972;3:257-260
- [Background] Nock MK, Park JM, Finn CT, Deliberto TL, Dour HJ, Banaji MR. Measuring the suicidal mind: implicit cognition predicts suicidal behavior. Psychol Sci. 2010 Apr;21(4):511-7. doi: 10.1177/0956797610364762. Epub 2010 Mar 9. PMID 20424092

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 participants were consented. Two were excluded for comorbid substance use disorder. 6 participants initiated treatment.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 8 participants were consented. 2 were excluded for comorbid substance use disorder. 6 initiated treatment.
Arm/Group | Cognitive Behavioral Therapy
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.50 (15.36)
Sex: Female, Male [Count of Participants; unit: Participants] — sex was self-reported
  Participants
    Female | 6
    Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Suicidal Ideation Intensity as Measured by the Columbia-Suicide Severity Rating Scale (C-SSRS) Intensity Subscale.
Description: The CSSRS intensity subscale measures frequency, duration, controllability, deterrents, and reasons for suicidal ideation. The scale ranges from 2-25 with higher scores indicating more severe suicidal ideation.
Time Frame: Pre-treatment, after treatment which was an average of 16 days, and through follow up, an average of 3 months post-treatment
Population: On participant was lost to follow-up and did not complete the 3 month follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre Cognitive Behavioral Therapy; Post Cognitive Behavioral Therapy; 3 Month Follow-up: Participants will receive up to 10 daily sessions of cognitive behavioral therapy (depending on length of stay), for about an hour each day. During this time the therapist will work to develop a crisis response plan and build coping skills to prevent future suicidal thoughts and behaviors.
  Cognitive Behavioral Therapy: Up to 10 daily sessions of brief cognitive behavioral therapy for suicidal inpatients for about an hour each day.
Arm/Group | Pre Cognitive Behavioral Therapy | Post Cognitive Behavioral Therapy | 3 Month Follow-up
Number analyzed (Participants) | 6 | 6 | 5
score on a scale | 13.0 (6.51) | 2.50 (6.12) | 2.60 (5.81)

2. Secondary Outcome: Structured Interview Guide for the Hamilton Rating Scale for Depression (SIGH-D)
Description: The SIGH-D is a clinician rated measure of depression symptom severity. Scores range from 0 to 52 with higher total scores indicating more severe depression.
Time Frame: Pre-treatment through post-treatment up to 24 days, 16 days on average
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pre Cognitive Behavioral Therapy | Post Cognitive Behavioral Therapy
Number analyzed (Participants) | 6 | 6
score on a scale | 15.0 (7.97) | 6.17 (3.60)

ADVERSE EVENTS:
Time Frame: Pre-treatment, after treatment up to 24 days, and through follow up, an average of 3 months post-treatment.
Groups:
- Cognitive-Behavioral Therapy: All participants received cognitive-behavioral therapy
Arm/Group | Cognitive-Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive-Behavioral Therapy (N=6)
vomiting (Gastrointestinal disorders) | 1 (1) — patient vomited during one of the CBT sessions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT03442699/Prot_SAP_000.pdf